CLINICAL TRIAL: NCT05580536
Title: Project Dulce for Arab Americans With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-7995
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Diabetes Self-Care; DSME; Genetic Education; Community Education; Arab Americans
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Project Dulce + Dulce Digital (Other): Participants will participate in a peer-led group diabetes self-management education and support program and receive ongoing support via text messages designed to improve knowledge, health beliefs, self-management behaviors and clinical outcomes.
  Interventions: Behavioral: Project Dulce + Dulce Digital

INTERVENTIONS:
Behavioral: Project Dulce + Dulce Digital — Project Dulce is a 5-week curriculum, group diabetes self-management education and support, program delivered by a peer educator in Arabic.
  The curriculum provides knowledge as well as skills and tools needed to change behaviors and adapt to a life with type 2 diabetes.
  The curriculum covers diabetes and its complication, the role of diet, exercise, and medication, and the importance of self-monitoring as well as the genetics contribution to diabetes development. It is presented over 5 weeks where participants will learn and practice diabetes self-management skills, and help one another address family, cultural, or health system barriers to managing their diabetes. .
  Following the 5-week curriculum, participants will be enrolled in the digital texting platform, Dulce Digital, in which they will receive on-going support via text messages derived from the curriculum, medication reminders, and blood glucose monitoring prompts in Arabic.

SUMMARY:
Arab Americans (AA) face many challenges in diabetes self-management due to the limited educational resources and support available for them. The cultural and linguistic barriers between patients and health care providers lead to poor diabetes management and outcomes. This study (Project Dulce Arabic) is adapted from the Project Dulce, an American Diabetes Association (ADA)-recognized Diabetes Self-Management Education Support (DSMES) program. Project Dulce Arabic comprises both peer-led diabetes education in Arabic and a 3-month text messaging program (Dulce Digital). The main aim of the study is to examine the effectiveness of a more culturally and linguistically appropriate diabetes education program in improving diabetes knowledge, beliefs, and self-management as well as hemoglobin A1C.

DETAILED DESCRIPTION:
Although the Arab American (AA) population is at a higher risk of pre-diabetes and type 2 diabetes (T2D) compared to the white non-Hispanic population, there are hardly any culturally appropriate diabetes self-management resources available for Arab Americans.

Project Dulce Arabic is a pilot study addressing both the linguistic and cultural barriers faced by the AA community in diabetes self-management while exploring the genetic background of type 2 diabetes in Arab Americans. To overcome the linguistic barriers, we adapt educational materials from the Project Dulce diabetes self-management study of Mexican Americans (A. Philis-Tsimikas et al., 2011). This 5-week peer-led educational program in Arabic aims to enhance type 2 diabetes knowledge, beliefs, and self-management behaviors as well as improving diabetes management measured by hemoglobin A1C after 3 months and 6 months in the study.

Project Dulce Arabic is incorporating genetic education as a part of its curriculum to raise the community awareness of the role of genetics in T2D development as well as the importance of early genetic risk detection for T2D prevention. We are also asking our Project Dulce Arabic participants to participate in the Scripps Bio-Repository (https://www.scripps.org/research/bio-repository). The specimens obtained from our study cohort will be used for genetic sequencing. Obtaining this genetic information will enable us to gain more insights into the genetic basis of type 2 diabetes in Arab Americans. Comparing the genetic risk of T2D, available from different biobanks, in other ethnic groups with that in Arab Americans would highlight the disease risk faced by the community and draw more attention towards the importance of early disease detection and prevention through tailored screening recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Are a participant of Metro Caring
* Self-identified Arab
* Diagnosed with type 2 diabetes mellitus (T2DM)
* HbA1c ≥7.5% in the last 30 days
* Able to speak, read, write, and comprehend in English and Arabic
* Have access to a cell phone that can receive/send text messages throughout the study

Exclusion Criteria:

* Pregnant
* Are currently participating in another diabetes-related study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Diabetes Knowledge at 3 months | 3 months
  Diabetes Knowledge Test (Diabetes Research and Training Center, University of Michigan, 2015) is a 23-item measure of diabetes knowledge, with general questions related to symptoms, self-management (e.g., diet, exercise, foot care, blood glucose monitoring, insulin), and complications (e.g., low, and high blood sugar). Greater scores indicate greater diabetes knowledge.
Change from Baseline Diabetes Knowledge at 6 months | 6 months
  Diabetes Knowledge Test (Diabetes Research and Training Center, University of Michigan, 2015) is a 23-item measure of diabetes knowledge, with general questions related to symptoms, self-management (e.g., diet, exercise, foot care, blood glucose monitoring, insulin), and complications (e.g., low, and high blood sugar). Greater scores indicate greater diabetes knowledge.
Change from Baseline Health Belief Model Scale at 3 months | 3 months
  Health Belief Model scale (Tan, 2004) is comprised of 36 items that evaluate the health beliefs and attitudes about complications prevention behaviors and active health related behaviors in individuals with diabetes. Responses are on a 5-point Likert-type scale (1=strongly disagree, 5=strongly agree), with lower scores indicating greater negative beliefs.
Change from Baseline Health Belief Model Scale at 6 months | 6 months
  Health Belief Model scale (Tan, 2004) is comprised of 36 items that evaluate the health beliefs and attitudes about complications prevention behaviors and active health related behaviors in individuals with diabetes. Responses are on a 5-point Likert-type scale (1=strongly disagree, 5=strongly agree), with lower scores indicating greater negative beliefs.
Change in Baseline Self-Efficacy for Diabetes Scale at 3 months | 3 months
  Stanford Self-Efficacy for Diabetes Scale (Lorig, Stewart, Ritter, et al., 1996) is comprised of 8 items that measure the confidence of a participant in performing self-care activities such as eating meals every 4 to 5 hours, following a healthful diet, exercising, and blood glucose monitoring. Response options range from 1=not at all confident to 10=totally confident, with higher scores indicating greater self-efficacy.
Change in Baseline Self-Efficacy for Diabetes Scale at 6 months | 6 months
  Stanford Self-Efficacy for Diabetes Scale (Lorig, Stewart, Ritter, et al., 1996) is comprised of 8 items that measure the confidence of a participant in performing self-care activities such as eating meals every 4 to 5 hours, following a healthful diet, exercising, and blood glucose monitoring. Response options range from 1=not at all confident to 10=totally confident, with higher scores indicating greater self-efficacy.
Understanding Health Implications of Genomics at 3 months | 3 months
  To assess the genetic knowledge, a 12-items questionnaire. Response options are 'agree', 'disagree', or 'don't know'. Similarly, a 13-items questionnaire with response options of 'agree' or 'disagree' will be used to assess the attitudes toward genetics research and testing.
Understanding Health Implications of Genomics at 6 months | 6 months
  To assess the genetic knowledge, a 12-item questionnaire. Response options are 'agree', 'disagree', or 'don't know'. Similarly, a 13-item questionnaire with response options of 'agree' or 'disagree' will be used to assess the attitudes toward genetics research and testing.

SECONDARY OUTCOMES:
Change in Baseline Summary of Diabetes Self-Care Activities at 3 months | 3 months
  Summary of Diabetes Self-Care Activities measure (Toobert, Hampson, & Glassgow, 2000) is a 13-item brief questionnaire that assesses a respondent's adherence to self-management behavior recommendations in the past 7 days, including general and specific diet, exercise, blood glucose testing, foot care, medication adherence, and smoking, with greater scores indicating greater adherence.
Change in Baseline Summary of Diabetes Self-Care Activities at 6 months | 6 months
  Summary of Diabetes Self-Care Activities measure (Toobert, Hampson, & Glassgow, 2000) is a 13-item brief questionnaire that assesses a respondent's adherence to self-management behavior recommendations in the past 7 days, including general and specific diet, exercise, blood glucose testing, foot care, medication adherence, and smoking, with greater scores indicating greater adherence.
Change in Baseline International Physical Activity Questionnaire-Short Form at 3 months | 3 months
  International Physical Activity -Short Form (Craig et al., 2003) assesses the amount of physical activity (work, leisure, and other) and sedentary time in the past 7 days.
Change in Baseline International Physical Activity Questionnaire-Short Form at 6 months | 6 months
  International Physical Activity -Short Form (Craig et al., 2003) assesses the amount of physical activity (work, leisure, and other) and sedentary time in the past 7 days.
Change in Baseline Food Frequency Questionnaire at 3 months | 3 months
  Food frequency questionnaire (Alqahtani et al., 2017) measures the amounts and frequencies of fruits, vegetables, and common foods in the Arab American community.
Change in Baseline Food Frequency Questionnaire at 6 months | 6 months
  Food frequency questionnaire (Alqahtani et al., 2017) measures the amounts and frequencies of fruits, vegetables, and common foods in the Arab American community.
Change in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 3 months | 3 months
  Samples will be processed by Quest Diagnostics Inc and assayed by Immunoturbidimetry (Integra 800, Roche).
Change in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 6 months | 6 months
  Samples will be processed by Quest Diagnostics Inc and assayed by Immunoturbidimetry (Integra 800, Roche).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khattab, MD, Principal Investigator — Scripps
Locations (2):
- United States (2):
  - San Ysidro Health, El Cajon, California
  - Metro Caring, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No